CLINICAL TRIAL: NCT04502940
Title: Can we Measure Pancreatitis Severity With Flow Cytometry?
Brief Title: Is Lymphocyte Subtype Important for Acute Pancreatitis Severity?
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Oguzkagan Batikan, Principal Investigator, Istanbul Training and Research Hospital
Other Study IDs: Pancreatitis 01.06.2020
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pancreatitis; Lymphocytic Infiltrate; Immune System Diseases
Keywords: pancreatitis; lymphocyte; Flow-cytometry
MeSH Terms: conditions — Pancreatitis; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild pancreatitis: Patients with mild acute biliary pancreatitis according to Atlanta classification
  Interventions: Diagnostic Test: Flow Cytometric analysis
- Moderate Pancreatitis: Patients with moderate acute biliary pancreatitis according to Atlanta classification
  Interventions: Diagnostic Test: Flow Cytometric analysis
- Severe pancreatitis: Patients with severe acute biliary pancreatitis according to Atlanta classification
  Interventions: Diagnostic Test: Flow Cytometric analysis
- Control: Healthy volunteers
  Interventions: Diagnostic Test: Flow Cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow Cytometric analysis — Blood samples will be taken from the patients with biliary pancreatitis and healthy volunteers to perform flow-cytometric analysis and to determine lymphocyte subgroups

SUMMARY:
Pancreatitis is a common complication especially in patients with gallbladder stones, most patients with biliary pancreatitis may recover spontaneously without sequelae, but in 10-20% of patients, the disease is severe and mortality rates of up to 30% are detected in these patients. In the evaluation of acute biliary pancreatitis, many scoring systems have been established (Atlanta, Ranson, APACHE, BISAP etc.) from past to present to determine morbidity and mortality of the disease.

In this study, the investigators aimed to evaluate the correlation between morbidity and mortality of acute biliary pancreatitis and lymphocyte subtypes with Flow-cytometry.

DETAILED DESCRIPTION:
Pancreatitis is a common complication especially in patients with gallbladder stones, most patients with biliary pancreatitis may recover spontaneously without sequelae, but in 10-20% of patients, the disease is severe and mortality rates of up to 30% are detected in these patients. In patients with severe pancreatitis, aggressive fluid replacement, organ damage follow-up, appropriate antibiotherapy, and endoscopic sphincterotomy and radiological interventions may be of great benefit. In the evaluation of acute biliary pancreatitis, many scoring systems have been established (Atlanta, Ranson, APACHE, BISAP etc.) from past to present to determine morbidity and mortality of the disease. There are limited number of studies in the literature about the immune parameters in the evaluation of acute pancreatitis. In a studies, serum inflammatory markers such as IL-1, IL-6 and CD4, CD8 T lymphocyte and Treg population were evaluated.Treg cells are reported to be an independent prognostic factor in determining the severity of acute pancreatitis. In patients diagnosed with acute biliary pancreatitis, determination of the course of the disease at the time of diagnosis is extremely important for treatment and survival.

In this study, the investigators aimed to evaluate the correlation between morbidity and mortality of acute biliary pancreatitis with lymphocyte subtypes via Flow-cytometry.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Diagnosis of acute biliary pancreatitis
* Sign the voluntary consent form

Exclusion Criteria:

* Being under 18 or older than 80
* Not signing the voluntary consent form
* Pancreatitis resulting from an interventional procedure (ERCP, surgery, etc.)
* Pregnant women
* Being a history of immunodeficiency
* Cancer history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Lymphocyte subtypes 1 | 9 months
  T helper (CD4) (%)
Lymphocyte subtypes 2 | 9 months
  T cytotoxic (CD8) (%)
Lymphocyte subtypes 3 | 9 months
  Treg (CD25 and CD127) (%)

CONTACTS AND LOCATIONS:
Overall Officials: Oguzhagan Batikan, M.D., Principal Investigator — İstanbul Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Training and Research Hospital, Istanbul
  - Gaziosmanpaşa Taksim Eğitim ve Araştırma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang W, Xiang HP, Wang HP, Zhu LX, Geng XP. CD4 + CD25 + CD127 high cells as a negative predictor of multiple organ failure in acute pancreatitis. World J Emerg Surg. 2017 Feb 2;12:7. doi: 10.1186/s13017-017-0116-7. eCollection 2017. PMID 28174597
- [Background] Yang Z, Zhang Y, Dong L, Yang C, Gou S, Yin T, Wu H, Wang C. The Reduction of Peripheral Blood CD4+ T Cell Indicates Persistent Organ Failure in Acute Pancreatitis. PLoS One. 2015 May 4;10(5):e0125529. doi: 10.1371/journal.pone.0125529. eCollection 2015. PMID 25938229
- [Background] Li J, Yang WJ, Huang LM, Tang CW. Immunomodulatory therapies for acute pancreatitis. World J Gastroenterol. 2014 Dec 7;20(45):16935-47. doi: 10.3748/wjg.v20.i45.16935. PMID 25493006